CLINICAL TRIAL: NCT03200249
Title: Preoperative Chemo-radiation With IG-IMRT Dose Escalation for Locally Advanced Rectal Cancers: Phase 2 Study (RADICAL)
Brief Title: Preoperative Chemo-radiation With IG-IMRT Dose Escalation for Locally Advanced Rectal Cancers
Acronym: RADICAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01083-48
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-01

CONDITIONS: Advanced Rectal Cancers
Keywords: dose escalation, chemo-radiation, rectum cancer, phase 2
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): 1. - Treatment : concomitant preoperative radio-chemotherapy (during 5 weeks)
     Chimiotherapy: Capecitabine 1600 mg/m2/j ; 5/7 days during the 5 weeks of radiotherapy
     Radiotherapy RT + SIB-IMRT (5 weeks ; 5 sessions/week ; 25 sessions): Pelvic prophylactic dose of 45 Gy (1,8 Gy/session); "boost" with a dose of 60 Gy on the tumor PTV (2,4 Gy/session) - Total dose: 60 Gy in 25 sessions during 5 weeks.
  2. - TME surgery (8 weeks after the end of treatment)
  Interventions: Radiation: Preoperative chemo-radiation with IG-IMRT dose escalation

INTERVENTIONS:
Radiation: Preoperative chemo-radiation with IG-IMRT dose escalation

SUMMARY:
Hypothesis : Therapeutic intensification by increasing the dose delivered to the tumor by RCMI (conformational radiotherapy by intensity modulation) in order to reduce local relapse, often associated with poor prognosis

Primary objective: evaluate the rate of tumor sterilization and the toxicities of RTCT with concomitant boost in intensity modulation in patients with rectal cancer CT3-T4 and / or cN1-2.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the rectum cT3 or cT4 or cN+, M0 and for which CPR recommends preoperative radiochemotherapy
2. Tumor <15 cm of the anal margin in rigid or subperitoneal rectoscopy at the MRI
3. Tumor potentially resectable from the outset, or considered to be resectable after radiochemotherapy
4. Operable Patient
5. Age between 18 and 75
6. OMS performance status 0-2
7. No co-morbidity likely to prevent the delivery of treatment
8. Adequate contraception for men, and for non-menopausal women
9. Neurotrophic neutrophils 1500 / mm3, platelets 100 000 / mm3, and hemoglobin 10 g / dL
10. Bilirubin ≤ 1.5 times the upper limit of normal (LNS), ASAT and ALAT ≤ 1.5LNS, Alkaline phosphatase ≤ 1.5 LNS
11. Creatinine clearance> 50 mL / min
12. Patient must have been informed and must have signed the specific informed consent form.
13. Patient must be affiliated to a Social Health Insurance.

Exclusion Criteria:

1. Remote metastasis
2. Cancer not resectable
3. Contraindication to capecitabine and its excipients
4. Previous history of pelvic radiotherapy or previous chemotherapy
5. History of inflammatory bowel or rectum disease
6. History of angina pectoris monitored or myocardial infarction or heart failure
7. Active active infection or other serious underlying condition that may prevent the patient from receiving treatment
8. Other concomitant cancer, or history of cancer other than in situ cancer of the treated cervix or basal cell carcinoma or squamous cell carcinoma
9. Patient already included in another therapeutic trial with an experimental molecule
10. Pregnant woman, likely to be pregnant or nursing
11. Persons deprived of their liberty or under guardianship
12. Patient unable to comply with the required medical follow-up for geographic, social or psychological reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Complete histological response rate | at 8 weeks after inclusion
  Absence of residual cancer cells on the final analysis of the tumor and lymph node

SECONDARY OUTCOMES:
Tolerance | at 1, 2, 3, 4, 5 and 13 weeks after inclusion and at 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months after surgery
  Toxicity is assessed according to the NCI-CTCAE toxicity scale version 4.0

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Besançon, Besançon
  - Centre Gf Leclerc, Dijon

IPD SHARING:
Plan to Share IPD: No